CLINICAL TRIAL: NCT00324493
Title: Musculoskeletal Function in Hemophilia in Developing Countries
Brief Title: Musculoskeletal Function in Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Other Study IDs: MUSFIH2004
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-06

CONDITIONS: Hemophilia
Keywords: Severe Hemophilia; Musculoskeletal Function; Factor Replacement
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Hemophilia, which results from deficiency of factor VIII or IX, is a common hereditary X-linked bleeding disorder affecting up to 10/100,000 population. About 60-70% of them have severe disease (factor level <1%). This group is characterized by the occurrence of frequent spontaneous bleeding into joints and soft tissues. If inadequately treated, it results in progressive damage to joints and muscles leading to crippling deformities. Close clinical observation of these patients over many years has shown that those with >1% levels have much less bleeding compared to those with less than 1%. This observation has gained immense clinical importance in planning therapy for these patients.

To prevent progressive joint damage, the missing factor needs to be replaced. Much has evolved in this practice in the last 50 years. From administration of whole blood in the beginning, to plasma and cryoprecipitate, to purified plasma-derived concentrates and finally recombinant factor concentrates. The standard of therapy now is to replace factors frequently enough to maintain >1% factor levels at all times ("prophylaxis") or administer immediately on premonition or earliest signs of bleeding ("on demand" therapy). This has greatly enhanced the quality of life of people with hemophilia. However, the optimal regimens of factor replacement remain to be defined. The definition of what is optimal management of this chronic condition, currently incurable for the vast majority of patients, varies significantly in different parts of the world, depending on practicality and social expectations. Models have care have been developed in Western countries based on careful documentation of outcome over many years. Such data is lacking from developing countries.

This multi-center study aims to systematically record the outcome of musculoskeletal function in people with hemophilia in developing countries for the first time and provide information that can help plan care for the 80% of all hemophiliacs in the world who live in these countries. Currently there is no well documented model of care at the range of factor replacement practiced in these countries nor is there any significant information on the long-term outcome of musculo-skeletal function among these patients.

DETAILED DESCRIPTION:
3.1 Musculoskeletal function in hemophilia - natural history

Severe hemophilia is characterized by recurrent bleeding into large joints and muscles resulting in progressive damage and deformity by the time the patient reaches the end of the second decade ultimately leading to severe functional disability in many of the affected people. This fact has been well known for long. The orthopedic outcome of a person with severe hemophilia was perhaps not very different in different parts of the world till the 1960s. However, in the last three decades, the ability of factor replacement therapy to completely modify the clinical outcome of severe hemophilia has been recognized. Factor replacement therapy itself has evolved much over this period and infusion of large quantities of factor concentrates has transformed the outlook of this condition. A person with hemophilia can now lead a nearly normal life without fear of frequent bleeding into joints.

3.2 Factor replacement for preserving musculoskeletal functions - the current models

As late as the early 1960s, factor replacement in large quantities was difficult because only fresh plasma could be used. With the discovery of cryoprecipitate in 1964, (1) larger quantities could be infused. Further purification and lyophilization made home-therapy possible. (2) It was soon obvious that early factor replacement could reduce joint damage significantly. Two schools of practice evolved: on-demand therapy where factor concentrates were infused at the earliest evidence of bleeding and prophylactic therapy aimed at maintaining factor level above 1% at all times. Both approaches required very large quantities of factor concentrates but could completely alter the expression of disease by preventing recurrent bleeding into joints. (3,4) What has facilitated this approach is the enhanced safety of plasma derived and recombinant factor concentrates. (5,6) Improved methods of donor selection and the introduction of viral inactivation steps in the manufacturing process have made these concentrates safer than ever before. (7)

The most convincing data on the effectiveness of prophylactic factor replacement in hemophilia is from Sweden. As shown with carefully documented long-term data, perfect joint architecture can be preserved with large quantities of factor concentrates ranging in doses from 4,000-9,000 IU/kg annually. (3) More recently, similar data from the Netherlands has shown that with much lower doses ranging from 1,400-2,500 IU/kg annually, joint damage can be very significantly reduced. (13) Unfortunately, both these studies have not reported the disability status of their patients in relationship to the extent of joint damage. In other words, it is not clear from this data whether the person with a joint score showing mild damage is necessarily worse functionally that someone with joint cores showing moderate damage. However, there is often a very large difference among them in terms of the total quantity of factor replacement therapy. In fact, clinical experience suggests that there is often a poor correlation between joint scores and functional disability in the joint. Optimal regimens for factor replacement therefore still remain to be defined. Two large multi-center studies to evaluate regimens for prophylactic therapy are underway in Italy and Canada.

3.3 Models for factor replacement in developing countries

While these models of replacement therapy are very effective in preventing arthropathy, they have also made hemophilia one of the most expensive diseases to treat. (8) Therefore the benefits of such an approach have been limited to those people with hemophilia who live in developed countries. (9) For three quarters of people with hemophilia in the world who live in developing countries, treatment of this nature remains a distant dream. Most of them receive very little or no factor concentrates. Blood bank products continue to be used for factor replacement therapy. (10) As efforts are made to improve their care, it is necessary to develop more practical models for management of hemophilia in these countries.

3.4 Aim of factor replacement therapy

The predominant cause of morbidity in hemophilia is the damage resulting from repeated bleeding into joints. It has therefore been the aim of therapy to establish a standard where there is no evidence of damage to the joints, clinically and radiologically. (11) The effectiveness of this approach in preserving joint integrity has been so good that it has now become the standard for therapy in economically developed countries. Unfortunately, the annual cost of such therapy at $50-100,000/person has been so high that it has been difficult even for countries with developed economies to adopt it universally.

It is certainly desirable for all people with hemophilia all over the world to have the same level of care. However, the reality is that it is simply not economically feasible. While the per capita GDP of developed economies are above $20,000, that of developing economies is in the range of $500-3,000. (12) Apart from this, attitude towards health care varies considerably with many countries spending less than $10 per person annually. In such situations, it is necessary to establish a different philosophy for factor replacement. The aim shifts from maintaining perfect joint integrity to reasonable joint function that will allow the person to remain functionally independent. Out of necessity and not out of choice, people with hemophilia in developing countries and their physicians have to accept this fact.

The situation with factor replacement for joint bleeding in developing countries is variable. The limited data available suggest that the total quantity of factor concentrate used varies from about 2-30,000 IU/person annually corresponding to about 25-500 iu/kg/year. (14,15) Some of these centers that use factor concentrates in the intermediate range have reported preservation of reasonable joint function and functional independence. However, this is not backed by carefully documented data on orthopedic outcome. A systematic evaluation of orthopedic outcome with the different replacement protocols will help develop suitable models for treatment of hemophilia in these countries and will also assist health care planners in determining the cost of care. In recent years, considerable efforts are being made in many developing countries to get support from governments or insurance agencies for hemophilia care but the absence of adequate data on outcome with protocols that are practical in these situations makes it difficult to convince the authorities that even lower doses can preserve long-term functional independence.

A unique aspect of this study will be the assessment of functional independence of people with hemophilia and its correlation with joint scores. Unfortunately assessment of functional independence measure in hemophilia has not been standardized. After much discussion at the WFH Congress at Seville and the subsequent meeting of the SSC of the ISTH with the prospective co-investigators and advisors, including Drs.Donna DiMichele, H. Marijke van den Berg, Bruce Evatt and Carol Kasper, it was decided to apply a generic instrument such as the WeeFIM® till a more hemophilia specific instrument becomes available. This instrument is easy to administer and has been shown to have excellent consistency. (16)

Baseline factor levels and quantum of factor replacement may not be the only determinants of musculo-skeletal outcome in hemophilia. Levels of other coagulation proteins, including presence of prothrombotic markers, can also alter clinical outcome. Polymorphisms of various modulators of the inflammatory response may play a role. Though it is not envisaged to study these parameters in this study, it has been planned to collect blood samples with informed consent for evaluating these some of these parameters in future, if possible.

Hypothesis While it is likely that there will be good correlation between joint scores and functional independence at low joint scores, this correlation is unlikely to be linear or even significant, with increasing joint scores.

This study aims to document the outcome of musculo-skeletal function in a large number of children with severe hemophilia receiving varying levels of factor replacement therapy over a long period of time with particular emphasis not only on joint scores but on the functional independence status of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia, defined as factor assay showing <1% activity (assay to be done using standard reagents), between 5-15 years of age
* Be willing to come for evaluation at least once in 6-12 months for 5 years

Exclusion Criteria:

* Detectable inhibitors by screening tests at recruitment

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250
Dates: Start 2004-06; Study Completion 2009-06

CONTACTS AND LOCATIONS:
Overall Officials: Alok Srivastava, MD, Principal Investigator — Christian Medical College, Vellore, India
Locations (10):
- Raul Perez Bianco, Buenos Aires, Buenos Aires F.D., Argentina
- Brazil (2):
  - Margareth Castro Ozelo /, Chagas, Cidade Univrsitaria Zeferino Vaz-Campinas-Sp
  - Elbio A.D' Amico / Jorge, São Paulo, São Paulo
- Magdy EI Ekiaby, Cairo, Cairo Governorate, Egypt
- Christian Medical College, Vellore, Tamil Nadu, India
- Mohammad Reza Baghaipour, Tehran, Tehran Province, Iran
- Tien Sim Leng, Singapore, Singapore
- Prof. Glynn Wessels, Tygerberg, South Africa
- Prof. Ampaiwan Chuansumrit, Bangkok, Thailand
- Norma De Bosch, Caracas, Venezuela